CLINICAL TRIAL: NCT04860921
Title: Oral Zinc Supplementation in Children With Dilated Cardiomyopathy : Aprospective Cohort Study in Assiut ,Egypt.
Brief Title: Zinc Deficiency in Dilated Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Abdel Hameed Ahmed, Principal investigator, Assiut University
Other Study IDs: Zinc in dilated cardiomyopathy
Record Dates: First submitted 2020-11-17; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Zinc Deficiency
Keywords: Dilated cardiomopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to detect effect of oral zinc supplementation in pediatric patients with dilated cardiomyopathy.

DETAILED DESCRIPTION:
Cardiomyopathies are group of heart diseases that influence cardiac muscles directly and are not related to hypertension, congenital, valvular and pericardial diseases. The most common type of cardiomyopathy is dilate cardiomyopathy.

Dilated cardiomyopathy usually manifests as chronic systolic heart failure leading to arrhythmias and sudden death.

Trace elements are known to have a key role in myocardial metabolism. The human heart requires energy from micro and macro nutrients both to regenerate proteins and cells, and to support cyclic contractions. Heart failure is associated with neuro-hormonal activation leading to elevated levels of inflammatory markers and oxidative stress.

Zinc is an essential micronutrient that impacts the cardiovascular system. There are multiple potential pathophysiologic causes for zinc deficiency in heart failure as result of impaired micronutrient consumption, hyper inflammatory state, diminished absorption and hyperzincuria from heart failure medications. Zinc deficiency may play a role as primary and possible reversible cause of dilated cardiomyopathy.

Plasma zinc levels have been reported in multiple observational studies of patients with heart failure particularly in studies of idiopathic dilated cardiomyopathy, serum zinc levels have been found to be low.

A small but growing body of evidence suggesting the role for oral zinc supplementation in the management of dilated cardiomyopathy however further evaluation of the impact on outcome is needed.

ELIGIBILITY:
Inclusion Criteria:

* children (1-18) year's age with impaired left ventricular systolic function due to dilated cardiomyopathy

Exclusion Criteria:

* patients with congenital heart diseases.
* patients less than one year age.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patiente between 1 and18 years with dilated cardiomypathy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-20 (Estimated); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
New york heart associaton functional classification for grading heart failure | 1.5 year
  All cases included the study will be carefully examined for sings of heart failure according to new york heart association classification for grading of heart failure

SECONDARY OUTCOMES:
Detailed echocardiographic examination | 1.5 year
  Detailed echocardiography using Phillips Envisor C according to the guidelines of the American society of echocardiography(18)،focusing on follow up of left ventricle end diastolic dimension Z-score ,left ventricle fractional shortening and ejection fraction.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maron BJ, Towbin JA, Thiene G, Antzelevitch C, Corrado D, Arnett D, Moss AJ, Seidman CE, Young JB; American Heart Association; Council on Clinical Cardiology, Heart Failure and Transplantation Committee; Quality of Care and Outcomes Research and Functional Genomics and Translational Biology Interdisciplinary Working Groups; Council on Epidemiology and Prevention. Contemporary definitions and classification of the cardiomyopathies: an American Heart Association Scientific Statement from the Council on Clinical Cardiology, Heart Failure and Transplantation Committee; Quality of Care and Outcomes Research and Functional Genomics and Translational Biology Interdisciplinary Working Groups; and Council on Epidemiology and Prevention. Circulation. 2006 Apr 11;113(14):1807-16. doi: 10.1161/CIRCULATIONAHA.106.174287. Epub 2006 Mar 27. PMID 16567565